CLINICAL TRIAL: NCT04324151
Title: Pembrolizumab Combined With Double Platinum Based Chemotherapy for Potentially Resectable Non-driver Gene Mutation Non-small Cell Lung Cancer
Brief Title: Pembrolizumab Combined With Double Platinum Based Chemotherapy for Potentially Resectable NSCLC
Status: Recruiting | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, professor, Hunan Province Tumor Hospital
Other Study IDs: PERSPECT
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the efficacy and safety of Pembrolizumab Combined With Double Platinum-Based Chemotherapy for Potentially Resectable Non-driver Gene Mutation Non-small Cell Lung Cancer

DETAILED DESCRIPTION:
Inclusion criteria:

diagnosed with Non-small cell lung cancer EGFR and ALK and ROS1 negative Treatment naive Potentially Resectable identified by MDT

ELIGIBILITY:
Inclusion Criteria:

* ≥18，Advanced Non-squamous Non-small Cell Lung Cancer Confirmed by Histopathology
* Potentially Resectable NSCLC
* Treatment Plan is Crizotinb or Standard Chemotherapy

Exclusion Criteria:

* Patients with contraindication of chemotherapy
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potentially Resectable Non-driver Gene Mutation Non-small Cell Lung Cancer
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2024-12-24 (Estimated); Study Completion 2025-03-24 (Estimated)

PRIMARY OUTCOMES:
PFS | may 2020- may 2021 (1 year)
  Progression free survival

SECONDARY OUTCOMES:
OS | may 2020- may 2021 (1 year)
  Overall survival
ORR | may 2020- may 2021 (1 year)
  To measure the patients's overall response rate

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China